CLINICAL TRIAL: NCT00222664
Title: Qidong Hepatitis B Intervention Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Qidong Liver Cancer Institute (Other); Merck Institute for Therapeutic Research (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Qidong-HBV-Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-08

CONDITIONS: Hepatitis B; Liver Neoplasms; Liver Diseases
Keywords: hepatitis B; hepatocellular carcinoma; prevention; vaccination
MeSH Terms: conditions — Hepatitis B; Liver Neoplasms; Liver Diseases; Carcinoma, Hepatocellular

INTERVENTIONS:
Biological: Hep-V Vax

SUMMARY:
During 1983-1990 in the Jiangsu province of China, 80,000 infants were randomised by area of birth between control, standard Hepatitis B vaccination (at 0, 1 and 6 months of age) and standard vaccination plus a booster dose at about 2 to 3 years of age. The aim is to prevent establishment of chronic HBV infection in early childhood, hence to prevent the morbidity of chronic hepatitis B in young adolescents and the incidence/mortality several decades later from liver cancer and other HBV related chronic liver diseases. Long-term follow-up through central registries will determine the impact of vaccination on liver cancer incidence and mortality.

ELIGIBILITY:
Inclusion Criteria:

all infants born in Qidong between September 1983 and November 1990

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 80000
Dates: Start 1983-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Zongtang Sun, MD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Richard Peto, Msc, Study Director — University of Oxford
Locations (3):
- China (2):
  - Qidong Liver Cancer Institute, Qidong, Jiangsu
  - Cancer Institute, Chinese Academy of Medical Sciences, Beijing
- Clinical Trial Service Unit and Epidemiological Studies Unit, Oxford, United Kingdom

REFERENCES:
- [Result] Sun Z, Zhu Y, Stjernsward J, Hilleman M, Collins R, Zhen Y, Hsia CC, Lu J, Huang F, Ni Z, et al. Design and compliance of HBV vaccination trial on newborns to prevent hepatocellular carcinoma and 5-year results of its pilot study. Cancer Detect Prev. 1991;15(4):313-8. PMID 1665400